CLINICAL TRIAL: NCT07020546
Title: Ovarian Platelet-Rich Plasma (oPRP) Injections Improvement In IVF Patients Based On Time-Lapse Incubator Culture for Automated Tracking and AI for Embryo Quality Assessment : A Non-Randomized Propsective Self-Controlled Interventional Study
Brief Title: Ovarian PRP Injections for Improved Embryo Quality Using Embryo Quality Score
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Generation Next Fertility (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IORG0010499-012025
Record Dates: First submitted 2025-05-13; First posted 2025-06-13 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Infertility; Poor Ovarian Reserve; Embryo Growth Disorder; in Vitro Fertilization
MeSH Terms: conditions — Infertility | interventions — Injections

STUDY DESIGN:
Intervention Model Description: A NON-RANDOMIZED PROSPECTIVE SELF-CONTROLLED INTERVENTIONAL STUDY
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Embryo Development Before and After Ovarian PRP Using Time-Lapse AI Embryo Quality Score (Experimental): Patients will undergo two IVF cycles. The first cycle will be before ovarian PRP treatment and the second will be after. The embryo development measured by data gathered in time-lapse imaging and AI software will be used to determine differences between the groups within the same patient
  Interventions: Procedure: Ovarian Platelet-rich plasma (PRP) injections

INTERVENTIONS:
Procedure: Ovarian Platelet-rich plasma (PRP) injections — This is a procedure that our patients receive at our clinic. We want to use the AI software to evaluate embryo development before and after treatment to see if there is a difference in embryo quality after PRP treatment within the same patient.

SUMMARY:
Patients will have ovarian PRP treatments and embryo development will be observed using time-lapse imaging and AI software.

DETAILED DESCRIPTION:
. oPRP Treatment & Second IVF Cycle (Study Cycle)

* Following the first IVF cycle, patients will undergo their first oPRP injection:

  * Timing: 1-2 weeks after the onset of the next menstrual cycle.
  * Procedure: Under IV sedation, a patient's autologous PRP will be prepared and injected directly into both ovaries under transvaginal ultrasound guidance.
* Second IVF Cycle (oPRP Study Cycle)

  * The same ovarian stimulation protocol will be used for consistency.
  * A second oPRP injection will be performed on stimulation days 2-5 to enhance folliculogenesis.
  * Ovulation will be triggered at the same follicular size thresholds, and oocyte retrieval will follow identical protocols.
  * Fertilization methodology will be identical to the first cycle unless no fertilization is identified in the first cycle.
  * Embryo Development Analysis: Up to 15 embryos will be cultured in the AI incubator, where time-lapse imaging will track their morphokinetics, and AI-based analysis will assess embryo viability and implantation potential.

ELIGIBILITY:
Inclusion Criteria:

* No none contraindications to IVF or PRP treatment
* Adequate ovarian reserves and AMH level
* Willingness to undergo two IVF cycles and oPRP treatment

Exclusion Criteria:

* Anovulation due to menopause or perimenopause
* Any health conditions that are contraindicated for IVF or oPRP treatment

Ages: 18 Years to 47 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-07-08 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Blastocyst formation and embryo quality | 1 year
  The number of high quality embryos that are created per cycle

SECONDARY OUTCOMES:
Live birth rate per transfer | 2 years
  The number of live births following embryo transfer

CONTACTS AND LOCATIONS:
Overall Officials: Jesse Hade, MD, Principal Investigator — Generation Next Fertility
Locations (1):
- Generation Next Fertility, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol (2025-06-01): https://cdn.clinicaltrials.gov/large-docs/46/NCT07020546/Prot_000.pdf
  • Informed Consent Form (2025-06-01): https://cdn.clinicaltrials.gov/large-docs/46/NCT07020546/ICF_001.pdf